CLINICAL TRIAL: NCT02292381
Title: Blood Flow Regulation in Glaucoma
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. Univ. Doz. Dr., Medical University of Vienna
Other Study IDs: OPHT-250313
Record Dates: First submitted 2013-10-22; First posted 2014-11-17 (Estimated); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Glaucoma Patients: Patients with primary open angle glaucoma
  Interventions: Other: Isometric exercise
- Healthy controls: age- and sex matched controls
  Interventions: Other: Isometric exercise

INTERVENTIONS:
Other: Isometric exercise

SUMMARY:
Glaucoma is one of the leading causes for blindness in industrialized countries. It is characterized by a progressive loss of retinal ganglion cells, morphological changes in the optic nerve head and a characteristic loss of visual field. Although increased intraocular pressure has been identified as the major risk factor for the development and the progression of the disease it has been speculated for a long time that impaired ocular blood flow may contribute to the pathogenesis of the disease. This concept has been supported by several epidemiological studies showing that low ocular perfusion pressure and small retinal vessel caliber are associated with the disease.

The proposed study tests the hypothesis that patients with glaucoma have reduced total retinal blood flow as compared to healthy subjects. Additionally, autoregulation of blood flow will be investigated during an increase in ocular perfusion pressure. This is of importance because it may clarify the degree of vascular involvement in glaucoma.

ELIGIBILITY:
Inclusion Criteria:

Patients with open angle glaucoma:

- Diagnosis of manifest open angle glaucoma as defined as pathological optic disc appearance, glaucoma hemifield test outside normal limits and/or untreated intraocular pressure ≥ 21 mmHg on at least three measurements in the medical history. Mean deviation in the visual field test < 10 decibel

Healthy control subjects:

* normal ophthalmic findings and intraocular pressure < 20 mmHg on at least three measurements
* no evidence of increased intraocular pressure in the medical history
* no signs of glaucomatous damage in the optic disc or the glaucoma hemifield test

Exclusion Criteria:

* Presence or history of a severe medical condition as judged by the investigator
* Abuse of alcoholic beverages
* Participation in a clinical trial in the 3 weeks preceding the study
* Exfoliation glaucoma
* Pigmentary glaucoma
* Secondary glaucoma
* Ocular hypertension
* History of acute angle closure
* Intraocular surgery within the last 6 months
* History of epilepsia
* Diabetes mellitus
* Ocular inflammation or infection within the last 3 months
* Untreated hypertension with systolic blood pressure >160 mmHg, diastolic blood pressure >95 mmHg
* Pregnancy or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 60 open angle glaucoma patients 60 healthy age- and sex matched controls
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2014-04 (Actual); Primary Completion 2016-11-28 (Actual); Study Completion 2016-11-28 (Actual)

PRIMARY OUTCOMES:
Optic nerve head blood flow | once

SECONDARY OUTCOMES:
Retinal blood flow | once

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria